CLINICAL TRIAL: NCT02202785
Title: A Phase 2 Trial of MLN0264 in Previously Treated Patients With Advanced or Metastatic Pancreatic Adenocarcinoma Expressing Guanylyl Cyclase C (GCC)
Brief Title: A Study of MLN0264 in Patients With Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision, No Safety or Efficacy Concerns
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C26003; 2014-000805-11 (EudraCT Number); U1111-1155-8964 (Other: WHO); REec-2014-1177 (Other: REec)
Record Dates: First submitted 2014-07-07; First posted 2014-07-29 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Drug therapy
MeSH Terms: interventions — indusatumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MLN0264 1.8 mg/kg (Experimental): MLN0264 1.8 mg/kg, 30-minute intravenous (IV) infusion, Day 1 of each 21-day cycle, for up to 1 year or until disease progression or unacceptable toxicity occurs (Up to 10 cycles). The dose may be decreased, delayed or discontinued in participants who develop treatment-associated nonhematologic and hematologic toxicity to MLN0264.
  Interventions: Drug: MLN0264

INTERVENTIONS:
Drug: MLN0264 — MLN0264 IV infusion

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of MLN0264 in patients with advanced or metastatic guanylyl cyclase C (GCC)-positive adenocarcinoma of the pancreas.

DETAILED DESCRIPTION:
The drug being tested in this study is called MLN0264. MLN0264 is being tested to treat tumors in people who have metastatic adenocarcinoma of the pancreas expressing guanylyl cyclase C (GCC). This study will assess tumor size reduction in patients who are administered MLN0264.

The study will enroll 42 to 81 patients. All participants will be administered MLN0264 at 1.8 mg/kg as a single, 30-minute, intravenous (IV) infusion on Day 1 of each 3-week treatment cycle, followed by a rest period of 20 days. Participants will continue to receive MLN0264 for up to 1 year or until disease progression or unacceptable toxicity occurs.

This multi-centre trial will be conducted worldwide. The overall time to participate in this study is approximately 19 months. Participants will make 3 to 6 visits to the clinic per treatment cycle, an end-of-treatment visit will occur 30 days after the last dose of study medication, and follow-up assessments will occur every 12 weeks until death or 6 months after the last patient completes treatment - whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years of age or older when written informed consent is obtained.
2. Histologically confirmed metastatic or advanced inoperable adenocarcinoma of the pancreas with immunohistochemistry (IHC) evidence of guanylyl cyclase C (GCC) expression indicated by an H-score of 10 or greater.
3. Treatment with 1 or more prior chemotherapies for advanced or metastatic adenocarcinoma of the pancreas.
4. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines. All scans and x-rays used to document measurable disease must be done within 28 days before enrollment (ascites and bone lesions are not considered measureable disease).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 14 days before enrollment.
6. Female participants who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 30 days after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)

   Male participants, even if surgically sterilized (ie, status postvasectomy), who:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.)
7. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
8. Adequate organ and hematological function as evidenced by the following laboratory values within 14 days before enrollment:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   * Platelet count ≥ 100 x 10^9/L
   * Hemoglobin ≥ 9 g/dL
   * Activated partial thromboplastin time (aPTT) ≤ 1.5 x the upper limit of the normal range (ULN) per institutional laboratory normal range
   * International normalized ratio (INR) ≤ 1.5 x ULN
   * Serum creatinine ≤ 1.5 x ULN
   * Total bilirubin ≤ 1.5 x ULN
   * Albumin ≥ 3g/dL
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
   * Serum lipase ≤ 3 x ULN and serum amylase within the normal range
9. Resolution of all toxic effects of prior treatments except alopecia to Grade 0 or 1 by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.
10. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Radiotherapy within 4 weeks before enrollment.
2. Concurrent treatment or treatment within 4 weeks of study entry with any other investigational agent or chemotherapy.
3. Female participants who are lactating and breastfeeding or have a positive pregnancy test during the Screening period.
4. Uncontrolled, clinically significant, symptomatic cardiovascular disease within 6 months before enrollment, including myocardial infarction, unstable angina, Grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication.
5. Treatment with any medication that has a clinically relevant potential risk of prolonging the QT interval or inducing torsades de pointes that cannot be discontinued or switched to a different medication before starting study drug.
6. Participants with electrocardiogram (ECG) abnormalities considered by the investigator to be clinically significant, or repeated baseline prolongation of the rate-corrected QT interval (QTc).
7. Ongoing or clinically significant active infection as judged by the investigator.
8. Signs of peripheral neuropathy (PN) ≥ NCI CTCAE Grade 2.
9. Concomitant chemotherapy, hormonal therapy, immunotherapy, or any other form of cancer treatment.
10. Use of strong cytochrome P450 (CYP) 3A4 inhibitors within 2 weeks before the first dose of study drug.
11. Any preexisting medical condition of sufficient severity to prevent full compliance with the study.
12. History of or current neoplasm other than gastric adenocarcinoma, except for curatively treated nonmelanoma skin cancer or in situ carcinoma of the cervix uteri.
13. Known diagnosis of human immunodeficiency virus (HIV) infection (testing is not mandatory).
14. Symptomatic brain metastases.
15. Ongoing anticoagulant therapy (eg, aspirin, coumadin, heparin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-07-02; Primary Completion 2016-01-15 (Actual); Study Completion 2016-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (16):
- United States (7):
  - Aurora, Colorado
  - St. Petersburg, Florida
  - Tampa, Florida
  - Boston, Massachusetts
  - Cincinnati, Ohio
  - Nashville, Tennessee
  - San Antonio, Texas
- Belgium (2):
  - Bruges
  - Leuven
- Spain (4):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Málaga, Malaga
  - Seville, Sevilla
- United Kingdom (3):
  - London, Greater London
  - Manchester, Greater Manchester
  - Sutton, Surrey

REFERENCES:
- [Derived] Almhanna K, Wright D, Mercade TM, Van Laethem JL, Gracian AC, Guillen-Ponce C, Faris J, Lopez CM, Hubner RA, Bendell J, Bols A, Feliu J, Starling N, Enzinger P, Mahalingham D, Messersmith W, Yang H, Fasanmade A, Danaee H, Kalebic T. A phase II study of antibody-drug conjugate, TAK-264 (MLN0264) in previously treated patients with advanced or metastatic pancreatic adenocarcinoma expressing guanylyl cyclase C. Invest New Drugs. 2017 Oct;35(5):634-641. doi: 10.1007/s10637-017-0473-9. Epub 2017 May 19. PMID 28527133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 26 investigative sites in Belgium, Spain, United Kingdom and the United States from 24 September 2014 to 15 January 2016.
Pre-assignment Details: Participants with a diagnosis of Pancreatic adenocarcinoma were enrolled in 1 treatment group, MLN0264 1.8 mg/kg, 30-minute IV infusion, Day 1 of each 21-day cycle.
Groups:
- MLN0264 1.8 mg/kg (GCC Low): MLN0264 1.8 mg/kg, 30-minute intravenous (IV) infusion, Day 1 of each 21-day cycle, for up to 1 year or until disease progression or unacceptable toxicity occurs (Up to 4 cycles). The dose may be decreased, delayed or discontinued in participants who develop treatment-associated nonhematologic and hematologic toxicity to MLN0264. Participants with guanylyl cyclase C (GCC) protein expression=Low (combined H-score 10-59). Total H-score 0-600 is the combined score of cytoplasmic staining 0-300 and apical staining 0-300 and is based on the percentage of tumor cells with staining intensity 1+, 2+ and 3+.
- MLN0264 1.8 mg/kg (GCC Intermediate): MLN0264 1.8 mg/kg, 30-minute IV infusion, Day 1 of each 21-day cycle, for up to 1 year or until disease progression or unacceptable toxicity occurs (Up to 10 cycles). The dose may be decreased, delayed or discontinued in participants who develop treatment-associated nonhematologic and hematologic toxicity to MLN0264. Participants with guanylyl cyclase C (GCC) protein expression=Intermediate (combined H-score 60-119). Total H-score 0-600 is the combined score of cytoplasmic staining 0-300 and apical staining 0-300 and is based on the percentage of tumor cells with staining intensity 1+, 2+ and 3+.
- MLN0264 1.8 mg/kg (GCC High): MLN0264 1.8 mg/kg, 30-minute IV infusion, Day 1 of each 21-day cycle, for up to 1 year or until disease progression or unacceptable toxicity occurs (Up to 6 cycles). The dose may be decreased, delayed or discontinued in participants who develop treatment-associated nonhematologic and hematologic toxicity to MLN0264. Participants with guanylyl cyclase C (GCC) protein expression=Intermediate (combined H-score >120). Total H-score 0-600 is the combined score of cytoplasmic staining 0-300 and apical staining 0-300 and is based on the percentage of tumor cells with staining intensity 1+, 2+ and 3+.
Period: Overall Study
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Started | 11 | 15 | 17
Completed | 0 | 0 | 0
Not Completed | 11 | 15 | 17
Not completed — Study Terminated by Sponsor | 1 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Reason not Specified | 10 | 7 | 13

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any amount of MLN0264.
Groups:
- Total: Total of all reporting groups
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High) | Total
Number analyzed (Participants) | 11 | 15 | 17 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (11.20) | 65.5 (7.41) | 62.9 (10.88) | 63.9 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 4 | 23
  Male | 3 | 4 | 13 | 20
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 9 | 15 | 17 | 41
  Black or African American | 1 | 0 | 0 | 1
  Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 8 | 14 | 17 | 39
Region of Enrollment [Number; unit: participants]
  Belgium | 1 | 4 | 0 | 5
  United States | 7 | 6 | 7 | 20
  United Kingdom | 1 | 1 | 1 | 3
  Spain | 2 | 4 | 9 | 15
Height [Mean (Standard Deviation); unit: cm] | 163.0 (13.20) | 162.1 (9.54) | 170.6 (8.51) | 165.7 (10.76)
Weight [Mean (Standard Deviation); unit: kg] | 60.98 (18.769) | 63.45 (18.465) | 71.20 (17.456) | 65.88 (18.261)
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.650 (0.3045) | 1.679 (0.2761) | 1.827 (0.2575) | 1.730 (0.2814)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors (RECIST)
Description: ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) as assessed by the investigator using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR: Disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.
Time Frame: Day 21, every other cycle, starting with Cycle 2 until disease progression, death or study closure (Up to 16 months)
Population: Response-Evaluable population included all participants with measurable disease who received at least 1 dose of MLN0264 and had at least 1 post-baseline response assessment.
Measure: Number; unit: percentage of participants
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 11 | 13 | 15
percentage of participants | 0 | 8 | 0

2. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Evaluation Findings
Description: Participants with at least one post-baseline potentially clinically significant serum chemistry, hematology, coagulation or urinalysis result. Clinically significant results are those that were assessed by the investigator to be Grade 3 or higher using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE). Grade 3=severe, Grade 4=life threatening or disabling and Grade 5=Death.
Time Frame: Day 1 of each 21 day cycle and 30 days after the last dose of study medication (Up to 7.9 months)
Population: Safety population included all participants who received any amount of MLN0264.
Measure: Number; unit: Participants
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 43
Participants
  Chemistry | 20
  Hematology | 16
  Coagulation | 23
  Urinalysis | 0

3. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Findings
Description: Participants with at least one potentially clinically significant post-baseline vital sign finding including measurements of diastolic and systolic blood pressure, heart rate, and oral temperature.
Time Frame: Day 1 of each 21 day cycle and 30 days after the last dose of study medication (Up to 7.9 months)
Population: Safety population included all participants who received any amount of MLN0264.
Measure: Number; unit: Participants
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 43
Participants | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time in days from the date of first study drug administration to the date of first documentation of disease progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Day 21 of every other 21-day cycle starting with Cycle 2, 30 days after the last dose of study medication, and then every 12 weeks for up to an additional 6 months (Up to 13.9 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 11 | 13 | 15
days | 39 [9 to 82] | 42 [21 to 218] | 41 [16 to 137]

5. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the date of first documentation of a Partial Response or better to the date of first documentation of disease progression or relapse based on investigator assessment using RECIST version 1.1 guidelines. Per RECIST version 1.1 for target lesions and assessed by MRI: CR, Disappearance of all target lesions; PR, >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: From first documented response until disease progression (Up to 16 months)
Population: Participants from the Response-Evaluable population, all participants with measurable disease who received at least 1 dose of MLN0264 and had at least 1 post-baseline response assessment, who had a response.
Measure: Median (Full Range); unit: days
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 1
days | 103 [103 to 103]

6. Secondary Outcome: Disease Control Rate
Description: Disease control rate is defined as the percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD) with a minimum of 12 weeks' duration. Investigator response is based on the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. CR: Disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum longest diameter (LD) since the treatment started.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 11 | 13 | 15
percentage of participants | 0 | 23 | 20

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time in days from the date of first study drug administration to the date of death.
Time Frame: Until death or 6 months after the last patient completes treatment-whichever occurs first (Up to 16 months)
Population: Safety population included all participants who received any amount of MLN0264.
Measure: Median (Full Range); unit: days
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 11 | 15 | 17
days | 162 [36 to 282] | 140 [43 to 443] | 162 [49 to 435]

8. Secondary Outcome: Cmax: Maximum Observed Serum Concentration for MLN0264
Time Frame: Cycles 1-3 predose and 10 minutes, 4 hours, and 3, 4, 8 and 15 days postdose. Cycles 4+ predose, 10 minutes, 4 hours, and 4 and 8 days postdose.
Population: Cmax was not a pre-specified secondary outcome measure. No data was collected.
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 0

9. Secondary Outcome: Serum Concentration of Monomethyl Auristatin E (MMAE)
Description: Blood samples were collected and sent to a laboratory to be tested for MMAE.
Time Frame: as for outcome 8
Population: PK-Evaluable population included all participants who received at least 1 dose of MLN0264 and who have sufficient MLN0264 concentration-time data to permit reliable estimation of MLN0264 exposure. "n" in the categories is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 43
ng/mL
  Cycle 1 Day 1, Pre-Dose | 0.000 (0.0000)
  Cycle 1 Day 1, 10 Minutes Post-Dose | 0.296 (0.1624)
  Cycle 1 Day 1, 4 Hours Post-Dose | 2.438 (1.3015)
  Cycle 1 Day 3, 48 Hours Post-Dose (n=41) | 5.205 (2.8110)
  Cycle 1 Day 4, 72 Hours Post-Dose (n=39) | 4.918 (2.3653)
  Cycle 1 Day 8, 168 Hours Post-Dose (n=43) | 2.994 (2.1173)
  Cycle 1 Day 15, 336 Hours Post-Dose (n=37) | 0.580 (0.5073)
  Cycle 2 Day 1, Pre-Dose (n=37) | 0.128 (0.1304)
  Cycle 2 Day 1, 10 Minutes Post-Dose (n=37) | 0.405 (0.3351)
  Cycle 2 Day 1, 4 Hours Post-Dose (n=37) | 2.665 (1.6053)
  Cycle 2 Day 3, 48 Hours Post-Dose (n=34) | 6.223 (3.5926)
  Cycle 2 Day 4, 72 Hours Post-Dose (n=32) | 5.808 (3.6296)
  Cycle 2 Day 8, 168 Hours Post-Dose (n=34) | 2.789 (2.0437)
  Cycle 2 Day 15, 336 Hours Post-Dose (n=28) | 0.560 (0.5332)
  Cycle 3 Day 1, Pre-Dose (n=9) | 0.145 (0.1318)
  Cycle 3 Day 1, 10 Minutes Post-Dose (n=9) | 0.395 (0.3514)
  Cycle 3 Day 1, 4 Hours Post-Dose (n=9) | 2.237 (1.6402)
  Cycle 3 Day 3, 48 Hours Post-Dose (n=8) | 6.563 (5.2034)
  Cycle 3 Day 4, 72 Hours Post-Dose (n=8) | 6.563 (6.2902)
  Cycle 3 Day 8, 168 Hours Post-Dose (n=7) | 2.826 (2.0234)
  Cycle 3 Day 15, 336 Hours Post-Dose (n=7) | 1.155 (1.2808)
  Cycle 4 Day 1, Pre-Dose (n=7) | 0.232 (0.2877)
  Cycle 4 Day 1, 10 Minutes Post-Dose (n=7) | 0.446 (0.4029)
  Cycle 5 Day 1, Pre-Dose (n=5) | 0.090 (0.0594)
  Cycle 5 Day 1, 10 Minutes Post-Dose (n=5) | 0.249 (0.1004)
  Cycle 6 Day 1, Pre-Dose (n=5) | 0.105 (0.0469)
  Cycle 6 Day 1, 10 Minutes Post-Dose (n=5) | 0.269 (0.1037)
  Cycle 6 Day 4, 72 Hours Post-Dose (n=5) | 4.234 (1.3134)
  Cycle 6 Day 8, 168 Hours Post-Dose (n=5) | 2.002 (0.9691)
  Cycle 7 Day 1, Pre-Dose (n=2) | 0.125 (0.0365)
  Cycle 7 Day 1, 10 Minutes Post-Dose (n=2) | 0.277 (0.0806)
  Cycle 8 Day 1, Pre-Dose (n=2) | 0.108 (0.0288)
  Cycle 8 Day 1, 10 Minute Post-Dose (n=2) | 0.257 (0.0481)
  Cycle 9 Day 1, Pre-Dose (n=2) | 0.050 (0.0179)
  Cycle 9 Day 1, 10 Minutes Post-Dose (n=2) | 0.190 (0.0361)
  Cycle 10 Day 1, Pre-Dose (n=1) | 0.132 (0.0000)
  Cycle 10 Day 1, 10 Minutes Post-Dose (n=1) | 0.385 (0.0000)
  End of Treatment (n=27) | 0.137 (0.1695)

10. Secondary Outcome: Guanylyl Cyclase C (GCC) H-score Assessed by Immunohistochemistry (IHC)
Description: GCC H-score is based on the sum of the 0 to 300 H-score for cytoplasmic staining and the 0 to 300 H-score for apical staining for a total possible H-score 0 to 600. Separate consent is required to obtain archival tumor specimens for GCC expression assessment prior to screening.
Time Frame: From pre-screening through end of study (approximately 18 months)
Population: Safety population included all participants who received any amount of MLN0264.
Measure: Mean (Full Range); unit: scores on a scale
Groups:
- MLN0264 1.8 mg/kg (GCC High): MLN0264 1.8 mg/kg, 30-minute IV infusion, Day 1 of each 21-day cycle,for up to 1 year or until disease progression or unacceptable toxicity occurs (Up to 6 cycles). The dose may be decreased, delayed or discontinued in participants who develop treatment-associated nonhematologic and hematologic toxicity to MLN0264. Participants with guanylyl cyclase C (GCC) protein expression=Intermediate (combined H-score >120). Total H-score 0-600 is the combined score of cytoplasmic staining 0-300 and apical staining 0-300 and is based on the percentage of tumor cells with staining intensity 1+, 2+ and 3+.
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 11 | 15 | 17
scores on a scale | 29.6 [10 to 55] | 84.0 [60 to 110] | 204.2 [120 to 355]

11. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An SAE is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event.
Time Frame: From the first dose through 30 days after the last dose of study medication (Up to 7.9 months)
Population: Safety population included all participants who received any amount of MLN0264.
Measure: Number; unit: Participants
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 11 | 15 | 17
Participants
  AEs | 11 | 15 | 17
  SAEs | 3 | 7 | 9

12. Secondary Outcome: MLN0264 Serum Concentrations
Description: Blood samples were collected and sent to a laboratory to be tested for serum concentrations of MLN0264.
Time Frame: as for outcome 8
Population: Pharmacokinetic (PK)-Evaluable population included all participants who received at least 1 dose of MLN0264 and who have sufficient MLN0264 concentration-time data to permit reliable estimation of MLN0264 exposure. "n" in the categories is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 43
μg/mL
  Cycle 1 Day 1, Pre-Dose | 0.000 (0.0000)
  Cycle 1 Day 1, 10 Minutes Post-Dose | 36.647 (10.0936)
  Cycle 1 Day 1, 4 Hours Post-Dose | 27.898 (8.4886)
  Cycle 1 Day 3, 48 Hours Post-Dose (n=41) | 6.950 (1.9173)
  Cycle 1 Day 4, 72 Hours Post-Dose (n=39) | 4.758 (1.5349)
  Cycle 1 Day 8, 168 Hours Post-Dose (n=43) | 1.563 (0.5818)
  Cycle 1 Day 15, 336 Hours Post-Dose (n=37) | 0.582 (0.2331)
  Cycle 2 Day 1, Pre-Dose (n=37) | 0.261 (0.1643)
  Cycle 2 Day 1, 10 Minutes Post-Dose (n=37) | 30.856 (9.9483)
  Cycle 2 Day 1, 4 Hours Post-Dose (n=37) | 26.691 (7.9664)
  Cycle 2 Day 3, 48 Hours Post-Dose (n=35) | 7.021 (2.4977)
  Cycle 2 Day 4, 72 Hours Post-Dose (n=32) | 4.432 (1.6115)
  Cycle 2 Day 8, 168 Hours Post-Dose (n=34) | 1.681 (0.7800)
  Cycle 2 Day 15, 336 Hours Post-Dose (n=27) | 0.692 (0.3038)
  Cycle 3 Day 1, Pre-Dose (n=9) | 0.431 (0.1481)
  Cycle 3 Day 1, 10 Minutes Post-Dose (n=9) | 34.978 (5.3350)
  Cycle 3 Day 1, 4 Hours Post-Dose (n=9) | 26.393 (3.3557)
  Cycle 3 Day 3, 48 Hours Post-Dose (n=8) | 9.486 (2.9593)
  Cycle 3 Day 4, 72 Hours Post-Dose (n=8) | 6.579 (1.8102)
  Cycle 3 Day 8, 168 Hours Post-Dose (n=7) | 1.701 (0.4201)
  Cycle 3 Day 15, 336 Hours Post-Dose (n=7) | 0.890 (0.2276)
  Cycle 4 Day 1, Pre-Dose (n=7) | 0.490 (0.1881)
  Cycle 4 Day 1, 10 Minutes Post-Dose (n=7) | 37.166 (9.3823)
  Cycle 5 Day 1, Pre-Dose (n=5) | 0.446 (0.2197)
  Cycle 5 Day 1, 10 Minutes Post-Dose (n=5) | 31.060 (8.3802)
  Cycle 6 Day 1, Pre-Dose (n=5) | 0.412 (0.2183)
  Cycle 6 Day 1, 10 Minutes Post-Dose (n=5) | 23.204 (12.9564)
  Cycle 6 Day 4, 72 Hours Post-Dose (n=5) | 4.689 (0.9286)
  Cycle 6 Day 8, 168 Hours Post-Dose (n=5) | 1.410 (0.2504)
  Cycle 7 Day 1, Pre-Dose (n=2) | 0.277 (0.0863)
  Cycle 7 Day 1, 10 Minutes Post-Dose (n=2) | 34.560 (6.5337)
  Cycle 8 Day 1, Pre-Dose (n=2) | 2.047 (2.6517)
  Cycle 8 Day 1, 10 Minute Post-Dose (n=2) | 27.120 (4.8649)
  Cycle 9 Day 1, Pre-Dose (n=2) | 0.178 (0.0467)
  Cycle 9 Day 1, 10 Minutes Post-Dose (n=2) | 31.880 (0.4808)
  Cycle 10 Day 1, Pre-Dose (n=1) | 0.207 (0.0000)
  Cycle 10 Day 1, 10 Minutes Post-Dose (n=1) | 20.860 (0.0000)
  End of Treatment (n=27) | 0.324 (0.2618)

13. Secondary Outcome: Serum Concentration of Total Antibodies (Conjugated and Unconjugated)
Description: Blood samples were collected and sent to a laboratory to be tested for conjugated and unconjugated antibodies.
Time Frame: as for outcome 8
Population: PK-Evaluable population included all participants who received at least 1 dose of MLN0264 and who have sufficient MLN0264 concentration-time data to permit reliable estimation of MLN0264 exposure."n" in the categories is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 43
μg/mL
  Cycle 1 Day 1, Pre-Dose | 0.000 (0.0000)
  Cycle 1 Day 1, 10 Minutes Post-Dose | 37.599 (9.4299)
  Cycle 1 Day 1, 4 Hours Post-Dose | 32.974 (8.1824)
  Cycle 1 Day 3, 48 Hours Post-Dose (n=41) | 14.051 (4.0368)
  Cycle 1 Day 4, 72 Hours Post-Dose (n=39) | 10.546 (3.6488)
  Cycle 1 Day 8, 168 Hours Post-Dose (n=43) | 5.252 (1.7703)
  Cycle 1 Day 15, 336 Hours Post-Dose (n=37) | 2.958 (1.1577)
  Cycle 2 Day 1, Pre-Dose (n=37) | 1.668 (0.7608)
  Cycle 2 Day 1, 10 Minutes Post-Dose (n=37) | 35.963 (10.9226)
  Cycle 2 Day 1, 4 Hours Post-Dose (n=37) | 32.134 (9.7822)
  Cycle 2 Day 3, 48 Hours Post-Dose (n=35) | 14.194 (4.8398)
  Cycle 2 Day 4, 72 Hours Post-Dose (n=32) | 10.948 (4.2741)
  Cycle 2 Day 8, 168 Hours Post-Dose (n=34) | 6.312 (2.7008)
  Cycle 2 Day 15, 336 Hours Post-Dose (n=27) | 3.923 (1.7465)
  Cycle 3 Day 1, Pre-Dose (n=9) | 2.654 (1.0757)
  Cycle 3 Day 1, 10 Minutes Post-Dose (n=9) | 39.500 (6.0580)
  Cycle 3 Day 1, 4 Hours Post-Dose (n=9) | 37.549 (8.2628)
  Cycle 3 Day 3, 48 Hours Post-Dose (n=8) | 19.181 (3.7260)
  Cycle 3 Day 4, 72 Hours Post-Dose (n=8) | 15.808 (2.0102)
  Cycle 3 Day 8, 168 Hours Post-Dose (n=7) | 6.631 (3.8091)
  Cycle 3 Day 15, 336 Hours Post-Dose (n=7) | 5.279 (1.9171)
  Cycle 4 Day 1, Pre-Dose (n=7) | 3.252 (1.3859)
  Cycle 4 Day 1, 10 Minutes Post-Dose (n=7) | 42.194 (8.8085)
  Cycle 5 Day 1, Pre-Dose (n=5) | 2.734 (1.2045)
  Cycle 5 Day 1, 10 Minutes Post-Dose (n=5) | 44.244 (27.1286)
  Cycle 6 Day 1, Pre-Dose (n=5) | 2.854 (1.7255)
  Cycle 6 Day 1, 10 Minutes Post-Dose (n=5) | 36.304 (12.1646)
  Cycle 6 Day 4, 72 Hours Post-Dose (n=5) | 12.667 (3.4384)
  Cycle 6 Day 8, 168 Hours Post-Dose (n=5) | 8.040 (3.1264)
  Cycle 7 Day 1, Pre-Dose (n=2) | 1.997 (0.7877)
  Cycle 7 Day 1, 10 Minutes Post-Dose (n=2) | 37.130 (4.9922)
  Cycle 8 Day 1, Pre-Dose (n=2) | 1.901 (0.5834)
  Cycle 8 Day 1, 10 Minute Post-Dose (n=2) | 66.240 (43.7558)
  Cycle 9 Day 1, Pre-Dose (n=2) | 1.462 (0.4547)
  Cycle 9 Day 1, 10 Minutes Post-Dose (n=2) | 34.790 (2.0789)
  Cycle 10 Day 1, Pre-Dose (n=1) | 1.282 (0.0000)
  Cycle 10 Day 1, 10 Minutes Post-Dose (n=1) | 26.320 (0.0000)
  End of Treatment (n=27) | 2.000 (1.2480)

14. Secondary Outcome: Percentage of Participants With Reduction From Baseline in Tumor Size
Description: The percentage of participants with the best percentage of tumor reduction from baseline in the sum of the diameter was calculated
Time Frame: Day 21 of each 21-day cycle, 30 days after the last dose of study medication, and then every 12 weeks for up to an additional 6 months (Approximately 13.9 months)
Population: Response-Evaluable Population was defined as all participants with measurable disease who receive at least 1 dose of MLN0264 and have at least 1 post-baseline response assessment.
Measure: Number; unit: percentage of participants
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 10 | 15 | 15
percentage of participants | 50 | 64 | 73

15. Secondary Outcome: Number of Participants With Antitherapeutic Antibodies (ATA)
Description: Blood samples were collected to assess the immunogenicity of MLN0264 (ATA development) using a laboratory test. Neutralizing ATA assessment was performed for ATA-positive samples only.
Time Frame: Pre-dose of each 21 day cycle and 30 days after last dose of study medication (Up to 7.9 months)
Population: Safety Population included all participant who received any amount of MLN0264.
Measure: Number; unit: Participants
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 11 | 15 | 17
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after the last dose of study drug (Up to 7.9 Months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- MLN0264 1.8 mg/kg: MLN0264 1.8 mg/kg, 30-minute IV infusion, Day 1 of each 21-day cycle, for up to 1 year or until disease progression or unacceptable toxicity occurs (Up to 10 cycles). The dose may be decreased, delayed or discontinued in participants who develop treatment-associated nonhematologic and hematologic toxicity to MLN0264.
Arm/Group | MLN0264 1.8 mg/kg
Serious Adverse Events (participants affected / at risk) | 19/43
Other Adverse Events (participants affected / at risk) | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN0264 1.8 mg/kg (N=43)
Intestinal obstruction (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1 — One treatment-emergent death occurred during treatment and is not related.
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1 — One treatment-emergent death occurred during treatment and is not related.
Bile duct obstruction (Hepatobiliary disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 — One treatment-emergent death occurred during treatment and is not related.
Device failure (General disorders) | 1
General physical health deterioration (General disorders) | 1 — One treatment-emergent death occurred during treatment and is not related.
Candida sepsis (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Biliary tract infection (Infections and infestations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MLN0264 1.8 mg/kg (N=43)
Anaemia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 19
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 11
Asthenia (General disorders) | 9
Fatigue (General disorders) | 16
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 4
Pyrexia (General disorders) | 6
Urinary tract infection (Infections and infestations) | 5
Blood alkaline phosphatase increased (Investigations) | 4
Weight decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 13
Dehydration (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 7
Headache (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 4
Dysuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.